CLINICAL TRIAL: NCT07197606
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Phase II Clinical Study to Evaluate the Efficacy and Safety of IxCell hUC-MSC-S in Patients With Ischemic Stroke in the Recovery Phase
Brief Title: Clinical Trial of Umbilical Cord Mesenchymal Stem Cells in Subacute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai IxCell Biotechnology Co., LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LC-MSC-IS25001
Record Dates: First submitted 2025-09-16; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSCs treatment (Experimental): Intravenous injection of mesenchymal stem cells
  Interventions: Drug: IxCell hUC-MSC-S (Human Umbilical Cord Mesenchymal Stem Cells)
- Placebo (Placebo Comparator): Intravenous injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Intravenous injection of placebo
  Arms: Placebo
Drug: IxCell hUC-MSC-S (Human Umbilical Cord Mesenchymal Stem Cells) — Intravenous injection of IxCell hUC-MSC-S
  Arms: MSCs treatment

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy, safety, and pharmacodynamic characteristics of Human Umbilical Cord Mesenchymal Stem Cells (hUC-MSCs) in adults with ischemic stroke in the anterior circulation during the recovery phase. Researchers will compare hUC-MSCs to a placebo to determine whether hUC-MSCs treatment is effective in treating recovery-phase anterior circulation ischemic stroke.

DETAILED DESCRIPTION:
This study aims to further evaluate the efficacy and safety of human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) in the treatment of stroke. Eligible participants will be randomized to receive either intravenous infusions of hUC-MSCs or a matching placebo. Over the 12-month study period, participants will be required to attend regular clinic visits for comprehensive neurological assessments, including the Fugl-Meyer Assessment (FMA), Modified Rankin Scale (mRS), National Institutes of Health Stroke Scale (NIHSS), Barthel Index (BI), and Mini-Mental State Examination (MMSE), as well as vascular imaging studies and biomarker analyses. Additionally, participants (or their caregivers, where applicable) will be instructed to consistently document neurological symptoms, functional activities, and the use of any rehabilitation medications or assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years, regardless of gender.
* 14 to 90 days after ischemic stroke.
* Clinical diagnosis of anterior circulation ischemic stroke.
* National Institutes of Health Stroke Scale (NIHSS) score is 6-20 points (inclusive), with NIHSS motor arm (item 5) or motor leg (item 6) score of 2-4 points, and NIHSS level of consciousness item (1a) score <2 points.
* It was anticipated that participants would either be able to give informed consent or have a legal representative who could do so.

Exclusion Criteria:

* People who had a history of epilepsy, dementia, Parkinson's disease, severe depression, or other neurological or psychiatric disorders.
* Intracranial hemorrhagic conditions.
* Pre-stroke mRS score >1.
* Severe cardiovascular disease.
* Severe pulmonary diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment motor score | 12 months
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based scale used to evaluate motor impairment. Its motor score, which ranges from 0 to 100, serves as a key parameter for quantifying motor recovery, where a higher score indicates better motor function.

SECONDARY OUTCOMES:
Modified Rankin Scale | 12 months
  The Modified Rankin Scale (mRS) is designed to evaluate the degree of dependence in daily activities rather than specific impairments. The mRS is a simple ordinal scale ranging from 0 to 6, where 0 indicates no symptoms and 6 indicates death. A lower score on the scale signifies a better level of independence and a lower degree of disability.
National Institutes of Health Stroke Scale | 12 months
  The National Institutes of Health Stroke Scale (NIHSS) is designed to evaluate the effects of a stroke on key functional domains such as consciousness, vision, motor strength, sensation, and language.The NIHSS score ranges from 0 to 42, with a higher score indicating more severe neurological deficits.
Barthel Index | 12 months
  The Barthel Index (BI) is commonly employed to evaluate functional disability and monitor rehabilitation progress in patients with chronic conditions or following events such as stroke. The total score ranges from 0 to 100, with a higher score indicating a greater degree of functional independence.
Mini-Mental State Examination | 12 months
  The Mini-Mental State Examination (MMSE) is a standardized screening tool designed to provide a quick assessment of an individual's global cognitive function.The total score ranges from 0 to 30, with a higher score indicating better cognitive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The general demographic data of participants, as well as clinical trial results including scoring data and safety data.
Supporting Information: Study Protocol
Time Frame: Individual Participant Data (IPD) is expected to be available upon trial completion on December 31, 2027, and this availability is anticipated to last until December 31, 2035.
Access Criteria: Relevant personnel who have submitted an application and obtained approval and authorization from the investigator(s) and sponsor(s) will receive the subjects' demographic data, scoring data, and safety data-with such information to be provided and transmitted by the investigator(s) to the authorized personnel.